CLINICAL TRIAL: NCT03264027
Title: A Multicenter Randomized Clinical Trial of Carbon Dioxide (CO2) Versus Air Insufflation for the Application of Argon Plasma to Reduce the Gastrojejunal Anastomosis in Individuals With Weight Regain After Bypass Surgery.
Brief Title: Carbon Dioxide Versus Air Insufflation for the Application of Argon Plasma to Reduce the Gastrojejunal Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Principal Investigator, Luiz Gustavo de Quadros, MD, MD, Kaiser Clinic and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kaiserargongjanastomosis
Record Dates: First submitted 2017-07-03; First posted 2017-08-28 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Dilatation of Anastomosis; Bypass Complication; Obesity
MeSH Terms: conditions — Obesity | interventions — Carbon Dioxide; Particulate Matter; Argon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the participant and the outcome assessor will be blinded to the study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon dioxide (Experimental): Argon fulguration will be performed using CO2 for insufflation. After using a disposable endoscopic catheter, argon plasma (Argon 2) (MAE, Ribeirão Preto, Brazil) will be applied in a 1-cm band around the entire circumference of the gastrojejunal anastomosis at an intensity of 90 W and a flow rate of 2 L/min.
  Interventions: Drug: Carbon dioxide; Drug: Argon fulguration
- Ambient air (Active Comparator): Argon fulguration will be performed using ambient air for insufflation. After using a disposable endoscopic catheter, argon plasma (Argon 2) (MAE, Ribeirão Preto, Brazil) will be applied in a 1-cm band around the entire circumference of the gastrojejunal anastomosis at an intensity of 90 W and a flow rate of 2 L/min.
  Interventions: Drug: Ambient air; Drug: Argon fulguration

INTERVENTIONS:
Drug: Carbon dioxide — Carbon dioxide will be used as an insufflating gas during argon fulguration of the dilatated anastomosis.
  Other Names: Carbon dioxide insufflation
  Arms: Carbon dioxide
Drug: Ambient air — Ambient air will be used as an insufflating gas during argon fulguration of the dilatated anastomosis.
  Other Names: Ambient air insuflattion
  Arms: Ambient air
Drug: Argon fulguration — The dilatated anastomosis from the gastric bypass surgery will be reduced in diameter using fulguration with argon. Patient in both groups will be placed in the left lateral decubitus position, with anesthesia being performed exclusively using propofol; adequate cardiopulmonary monitoring will be carried out during the entire procedure. After sedation, endoscopy will be performed with an Olympus CV-180 endoscope (Olympus, Tokyo, Japan) and analysis and measurement of the anastomosis will be achieved using Raptor foreign body forceps (Endoscopy Group US, Inc., Mentor - Ohio, USA). The images will be transferred to an Olympus EvisExera II processor connected to a computer with the ZScan 5 program (Goiânia, GO, Brazil).
  Other Names: Argon

SUMMARY:
The objective of this randomized clinical trial is to compare pain levels during and after insufflation with carbon dioxide or in subjects that will undergo endoscopic fulguration with argon to reduce the diameter of the gastrojejunal anastomosis. The investigators hypothesize that carbon dioxide will be superior in causing less pain and leading to less discomfort.

DETAILED DESCRIPTION:
Laparoscopic gastric bypass surgery is one of the strategies oriented towards weight reduction in obese patients. Although in the short term it has a high degree of success, weight regain is common in the long term, in part due to the dilatation of the anastomosis that allows food to pass without barriers and hinders the purpose of bypass surgery. Fulguration with argon is an endoscopic technique that reduces the diameter of the anastomosis, offering resistance to food passage and improving patient outcomes.

Although carbon dioxide is the current standard for laparoscopic surgery, its use for fulguration with argon as compared to ambient air has not been investigated in the setting of the stenosis of a dilated anastomosis following gastric bypass surgery. stenosis. Therefore, to investigate pain during and after this procedure, investigators will conduct a randomized clinical trial comparing carbon dioxide and ambient air.

The secondary aims will be to measure the diameter of the gastrojejunal anastomosis during three endoscopic sessions and in a final control examination eight weeks after the third session; to determine whether the patient loses weight or not by the final control objective after three sessions of endoscopic fulguration with argon; to analyze if the method employed is able to reduce body weight to the minimum weight achieved after bariatric surgery;and to investigate whether there is a correlation between the percentage reduction in anastomotic diameter and the percentage loss of regained weight.

ELIGIBILITY:
Inclusion Criteria:

* Regain of at least 10.0% of the minimum weight reached after the gastric bypass;
* Ability to understand study procedures;
* Signed the informed written consent form;
* Possible to complete all the stages of the study.

Exclusion Criteria:

* Presence of very tight restrictive ring preventing the advancement of the endoscopy device;
* Stenosis of the anastomosis preventing the progression of the endoscopy device before the end of the three endoscopic sessions;
* History of liver diseases such as cirrhosis or chronic active hepatitis;
* Patients who required anticoagulant therapy with the exception of antiplatelet agents;
* Pregnant women or those intending to become pregnant within 12 months after fulguration with argon;
* Participant in another ongoing clinical research;
* Recent history of neoplasia (less than 5 years);
* Alcoholism or drug use;
* HIV positive;
* Unbalanced or uncontrollable psychiatric disorders;
* Anemia or severe nutritional deficiencies;
* Allergy to anesthetic compounds;
* Impossibility to return within defined periods for consultations and endoscopic sessions of fulguration with argon;
* Inability to follow nutritional guidelines after each endoscopic session;
* Inability to understand study procedures;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain Visual Analogue Scale | Before surgery, and after eight weeks of the first endoscopic session. The outcome will be the substraction of the initial value and the final value of pain.
  A visual scale to assess self-reported pain going from 0 to 10.

SECONDARY OUTCOMES:
Change in diameter of the gastrojejunal anastomosis | Before surgery, and after eight weeks of the first endoscopic session.
  Analysis and measurement in millimeters of the anastomosis will be achieved using Raptor foreign body forceps (Endoscopy Group US, Inc., Mentor - Ohio, USA).
Weight reduction | Before surgery, and after eight weeks of the first endoscopic session.
  The final weight measured in kilograms after eight weeks of the initial surgery will be subtracted from the weight at the start of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Luiz G Quadros, MD, Principal Investigator — Kaiser Clinic and Hospital
Locations (1):
- Kaiser Clinic and Day Hospital, São José Do Rio Prêto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baretta GA, Alhinho HC, Matias JE, Marchesini JB, de Lima JH, Empinotti C, Campos JM. Argon plasma coagulation of gastrojejunal anastomosis for weight regain after gastric bypass. Obes Surg. 2015 Jan;25(1):72-9. doi: 10.1007/s11695-014-1363-2. PMID 25005812